CLINICAL TRIAL: NCT03832348
Title: 18-FDG Tumour Metabolism Changes in PDL1 Superior to 50% Stage III/IV Non Small Cell Lung Cancer During First Line Treatment With Pembrolizumab
Brief Title: Dynamics of 18-FDG Uptake in Stage III/IV Non Small Cell Lung Cancer During First Line Pembrolizumab Treatment
Acronym: iTEP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB18.05
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: PET scan imaging; Pembrolizumab; Response; Parametric imaging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET scan imaging (Experimental): PET scan will be performed each of three first cycles of pembrolizumab to describe the early tumour metabolic changes during the first line of treatment.
  Interventions: Device: PET scan imaging

INTERVENTIONS:
Device: PET scan imaging — 3 PET scans will be performed after each 3 first infusions of Pembrolizumab

SUMMARY:
The aim of this study is to describe the early dynamics of 18-FDG uptake in non smal cell lung cancer during first line treatment with pembrolizumab, and to evaluate whether or not they differ according to treatment response at 3 months.

DETAILED DESCRIPTION:
Immunotherapy with anti-PD1 antibody, such as Pembrolizumab, is widely used in the treatment of stage III/IV non small cell lung cancer. In order to refine treatments and patients' prognosis, early assessment of tumour response is needed.

The aim of this study is to describe the early tumour metabolic changes in non smal cell lung cancer during first line treatment with pembrolizumab, and to evaluate whether or not they differ according to treatment response.

Eligible patients with stage III/IV, PDL1>50% NSCLC will receive pembrolizumab treatment as per standard of care.

Tumour metabolism will be assessed by 18-FDG PETscan before each of the 3 first pembrolizumab infusions. Treatment response will be determined by RECIST, irRC and mCHOI criteria at 3 months.

Prognostic and predictive value of baseline and dynamic metabolic parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Non operable non small cell lung cancer
* Indication of treatment by Pembrolizumab
* PD-L1 status superior to 50 %
* Age more than 18 years
* At least one measurable target
* Written inform consent

Exclusion Criteria:

* no treatment by pembrolizumab
* immunosuppressive treatment
* uncontrolled diabete
* Pregnancy or breast-feeding
* curatorship or guardianship
* not possibility to follow-up the procedures of the study due to geographic, social or psychic reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Determination of progression by early PET scan | 3 months
  Determination of non-response of treatment by PET scan imaging after one cycle of Pembrolizumab

SECONDARY OUTCOMES:
Progression free survival | 24 months
  Time between inclusion and progression
Overall survival | 24 months
  Time between inclusion and death

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Becker, MD, Principal Investigator — Centre Henri Becquerel; Florian Guisier, MD, Principal Investigator — CHU Rouen
Locations (2):
- France (2):
  - Centre Henri Becquerel, Rouen
  - CHU, Rouen